CLINICAL TRIAL: NCT06446778
Title: Pipeline Embolization Device for Intracranial Aneurysm (PEDIA): a Prospective, Multicenter Cohort Focus on Safety, Efficacy, and Haemodynamics
Brief Title: Pipeline Embolization for Intracranial Aneurysms
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); Zhongshan Hospital Of Traditional Chinese Medicine (Other); First Affiliated Hospital of Jinan University (Other); Beijing Tiantan Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Affiliated Hospital of Southwest Medical University (Other); Guangdong 999 Brain Hospital (Other); Shantou Central Hospital (Other); Guangdong Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: LC2024ZD027
Record Dates: First submitted 2024-05-22; First posted 2024-06-06 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Efficacy, Self; Hemodynamic Instability; Stenosis; Aneurysm, Intracranial
Keywords: intracranial aneurysms; flow-diverter device; Pipeline embolization device; in-stent stenosis
MeSH Terms: conditions — Constriction, Pathologic; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Saccular aneurysms: Patients with saccular aneurysms were enrolled.
  Interventions: Device: Pipeline embolization device with or without shield technique
- Non-saccular aneurysms: Patients with non-saccular (i.e., fusiform, dissecting, blood blister-like) aneurysms were enrolled.
  Interventions: Device: Pipeline embolization device with or without shield technique

INTERVENTIONS:
Device: Pipeline embolization device with or without shield technique — The patients undenwent Pipeline embolization device implantation with or without shield technique due to market availability, choice and preferences of the surgeon.

SUMMARY:
This study collected the clinical, laboratory, and imaging data from patients with intracranial aneurysms, who underwent Pipeline implantation. The purpose of this study is to observe the safety, effcacy, and haemodynamics after Pipeline embolization.

DETAILED DESCRIPTION:
This study collected the clinical, laboratory, and imaging data from patients with intracranial aneurysms, who underwent Pipeline implantation. The purpose of this study is to observe the safety, effcacy, and haemodynamics after Pipeline embolization. The primary outcomes were aneurysmal occlusion status, incidence of in-stent stenosis, and functional prognosis. The secondary outcomes were hemodynamic changes before and after stent implantation.

ELIGIBILITY:
Inclusion criteria:

1. Aged 22 to 75 years old, male or non-pregnant female;
2. UIA was diagnosed by CTA, MRA, or DSA;
3. The size of aneurysms is between 3 to 25mm;
4. Understands the nature of the procedure and provision of written informed consent;
5. Indications for FD implantation with or without adjunctive coiling;
6. Is willing to return to the investigational site for follow-up according to our protocol.

Exclusion criteria:

1. With contraindications to flow-diversion treatment or known allergy to cobalt-chromium alloy or contrast medium;
2. Pregnancy or lactation;
3. Coexist with other vascular lesions (coronary artery disease, abdominal aortic aneurysm, severe intracranial artery stenosis, arteriovenous malformation, dural arteriovenous fistula, Moyamoya disease, etc.);
4. Parent vessel with a diameter <2.0 mm or ≥5.0 mm.;
5. Unwilling to be followed up or likely to have poor treatment compliance;
6. Life expectancy less than 3 years;
7. Inability to receive anti-platelet or anticoagulant medication;
8. Severe neurological deficit that renders the patient unable to live independently (modified Rankin score ≥4);
9. Enrollment in another trial or other situations that the researcher deems unsuitable for inclusion in the study.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent Pipeline implantation for intracranial aneurysms
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
The occlusion rate of the aneurysm | 1 years
  The occlusion rate of the aneurysm at 6 months；O'Kelly Marotta classification: complete occlusion (D, entirely non-filling), near-complete occlusion (C, only entry remnant), and incomplete occlusion (A and B, subtotal and total filling).

SECONDARY OUTCOMES:
in-stent stenosis | 1 years
  In-stent stenosis is defined as a growth process beyond the limits of stent mesh, which appears as a visible gap between the vessel lumen filled with contrast agent and stent struts.
  Stenosis ratio (SR) = [1-(actual diameter of the most stenotic segment with digital subtraction/actual diameter of stent measured on without digital subtraction)]*100%
  When there was no appreciable gap, cases were described as patency. Intimal hyperplasia was labeled when the SR was less than 25 %. ISS was defined as an SR of ≥ 25 %, and the stenosis grade was classified as mild (25 % to 49 %), severe (50 % to 99 %), or lumen occlusion (SR = 100 %)
perioperative complications | 1 months
  perioperative complications；such as arterial perforation, iatrogenic arterial dissection, embolization in previously uninvolved vascular territory, arterial access site hematoma, and retroperitoneal hematoma. Arterial perforation will be defined at angiography by the operator and associated with subarachnoid hemorrhage. Iatrogenic arterial dissection will be defined at angiography by the operator. Arterial access site hematoma will be assessed as a complication of arterial access puncture and defined by clinical examination and anatomic imaging. Retroperitoneal hematoma will be assessed as a complication of groin puncture and defined by imaging (ultrasound or CT or MR angiography). The definition of embolization in previously uninvolved vascular territory is noted after recanalization of the primary occlusion site, any vessel occlusions distal from the primary occlusion site are considered emboli due to periprocedural thrombus fragmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanzhi Duan, MD, Study Director — Zhujiang Hospital
Locations (1):
- Zhujiang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Huang C, Zhu Y, Feng X, Tong X, Wen Z, Lin J, Huang M, Yuan H, Dai L, Chen W, Hu Y, Bi Y, Deng X, Xie Z, Shang G, Luo Y, Zhao Y, Peng C, Huang C, Su S, Zhang X, Li X, Guo Z, Liu A, Duan C. Stent match of pipeline embolization device: prediction of incomplete occlusion and in-stent stenosis by actual stent size after implantation. Neurosurg Rev. 2025 May 30;48(1):462. doi: 10.1007/s10143-025-03625-8. PMID 40442402
- [Derived] Huang J, Huang Y, Feng X, Huang C, Huang M, Wen Z, Xu A, Ge R, Yuan H, Shi H, Ma G, Li C, Lin J, Yi R, Hu Y, Jin Y, Liang S, Bi Y, Su S, Zhang X, Li X, Duan C. Predictive value of the systemic immune-inflammation index for periprocedural complications in flow diverter treatment for patients with intracranial aneurysms. Neurosurg Rev. 2024 Oct 22;47(1):809. doi: 10.1007/s10143-024-03053-0. PMID 39436476